CLINICAL TRIAL: NCT06404125
Title: Investigation of the Effect of Pre-treatment Central Sensitization Severity on Steroid Injection Results in Rotator Cuff-induced Shoulder Pain
Brief Title: Investigation of the Effect of Central Sensitization Symptom Severity on Steroid Injection Results in Shoulder Pain
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 23/20
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Rotator Cuff Lesion; Subacromial Impingement Syndrome; Shoulder Pain; Chronic Pain
Keywords: central sensitization; chronic pain; Subacromial; Shoulder; Pressure
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (Patients without central sensitization): Patients with rotator cuff lesions lasting more than three months and without central sensitization will be included in group 1. (n=18)
  Interventions: Diagnostic Test: Range of Motion of Shoulde Joint; Diagnostic Test: Hand Grip Test; Diagnostic Test: Numeric Rating Scale; Diagnostic Test: Pain-Pressure Threshold Measurement With an Algometer; Diagnostic Test: Quick Disabilities of the Arm, Shoulder and Hand (Quick-DASH); Diagnostic Test: Short Form-36; Diagnostic Test: Central Sensitization Scale; Diagnostic Test: Hospital Anxiety and Depression Scale
- Group 2 (Patients with central sensitization): patients with rotator cuff lesions lasting more than three months and central sensitization will be included in group 2. (n=18)
  Interventions: Diagnostic Test: Range of Motion of Shoulde Joint; Diagnostic Test: Hand Grip Test; Diagnostic Test: Numeric Rating Scale; Diagnostic Test: Pain-Pressure Threshold Measurement With an Algometer; Diagnostic Test: Quick Disabilities of the Arm, Shoulder and Hand (Quick-DASH); Diagnostic Test: Short Form-36; Diagnostic Test: Central Sensitization Scale; Diagnostic Test: Hospital Anxiety and Depression Scale

INTERVENTIONS:
Diagnostic Test: Range of Motion of Shoulde Joint — Goniometric measurements will be made for both upper extremities. Flexion, extension, abduction, adduction, internal and external rotation angles of the shoulder complex will be evaluated in the measurement.
Diagnostic Test: Hand Grip Test — The purpose of this test is to test the maximum isometric contraction strength of the hand and forearm muscles. A hand grip dynamometer (Jamar) will be used for the test. While the patient is sitting in the chair, the elbows will be close to the body and at 90 degree flexion, the wrist will be in a neutral position. The patient will be asked to grasp the dynamometer and squeeze it as hard as she can, and the average of 3 measurements made with an interval of 10 seconds. The test will be repeated for both upper extremities separately.
Diagnostic Test: Numeric Rating Scale — Shoulder pain, feeling of tension and heaviness on the affected arm will be evaluated separately by numerical scale.
Diagnostic Test: Pain-Pressure Threshold Measurement With an Algometer — The measurement will be performed 2 times with 3 min intervals for each region and the average of these applications will be recorded. Before the test, a trial test will be applied to the patient. With the pressure algometer, pressure will be applied to the selected points until it causes pain and the test will be terminated for that region when the patient feels pain.
  The measurement includes bilateral shoulder region and left forearm as control region and Wagner manual pressure algometer (1 cm2 probe-10 kg/20 lb) will be used. The selected points will be:
  1. Bilateral supraspinatus muscle: 1 cm cranial to the midpoint of the spina scapulae
  2. Bilateral infraspinatus muscle: Medial edge of the scapula, intersection of the spina scapula and the inferior scapular angle
  3. Bilateral upper trapezius muscle: MidN point of the line joining the acromion and C7 spinous process
  4. Left forearm volar face center as control point
Diagnostic Test: Quick Disabilities of the Arm, Shoulder and Hand (Quick-DASH) — The arm, shoulder and hand problems rapid questionnaire is a shortened version of a questionnaire designed to detect symptoms and loss of function secondary to musculoskeletal problems of the upper extremity. The questionnaire will be used to assess quality of life related to upper extremity function.
Diagnostic Test: Short Form-36 — The scale was developed by Ware in 1987 and consists of 36 questions in which 8 sub-parameters related to the health status of the person are questioned. These parameters are physical function, pain, limitation due to physical and emotional problems, emotional well-being, social function, fatigue and general health perception. The Turkish validity and reliability of the scale was performed by Pınar et al. It is one of the leading methods used in the evaluation of quality of life in our country as well as all over the world.
Diagnostic Test: Central Sensitization Scale — The central sensitization scale was developed primarily to detect central sensitization findings in patients with chronic pain and consists of two parts, A and B. In part A, 25 somatic and psychosocial symptoms frequently found in patients with central sensitization are questioned. In part B, the presence of diseases with a well-defined relationship with central sensitization is questioned without participating in the scoring. Patients who score 40 points or more out of a total of 100 points are considered to have central sensitization. Düzce et al. stated that the Central Sensitization Scale can be used as a valid method in the Turkish population to screen the presence of central sensitization in patients presenting with chronic pain.
Diagnostic Test: Hospital Anxiety and Depression Scale — This scale was developed by Zigmond and Snaith in 1983 to screen anxiety and depression in individuals with physical illness. The scale consists of fourteen questions, seven for anxiety and seven for depression, to be answered on a four-point Likert scale. The Turkish validity and reliability of the scale has been demonstrated and a score above ten for anxiety and seven for depression is considered significant.

SUMMARY:
The aim of this study was to investigate the effect of the presence and severity of pre-treatment central sensitization on the results of subacromial/ intra-articular shoulder injection in patients with rotator cuff lesion/subacromial impingement. The hypothesis of the study is that the treatment response will decrease in patients with pre-injection central sensitization.

There are many studies investigating the frequency of central sensitization in various shoulder pathologies. However, the effect of this condition, which is likely to be associated with chronic pain in these patients, on treatment response is unknown. The effect on the results of shoulder injection, one of the most common procedures in physical therapy practice, will be investigated.

DETAILED DESCRIPTION:
Shoulder pain is one of the most common musculoskeletal complaints and its prevalence varies between 7-26%. Although some of the patients with shoulder pain show complete recovery, pain persists in some of them. One of the most common sources of pain in these patients is subacromial impingement syndrome (SIS) leading to rotator cuff pathology. The multifactorial nature of pain in these patients makes the treatment of SIS difficult.

Central sensitization (CS) has been reported as one of the factors associated with persistence of pain in patients with shoulder pain in different etiologies, especially in the SIS. CS can be summarized as an increase in the response of neurons located in the central nervous system to subthreshold stimuli and is the source of chronic pain in many diseases. A decrease in the pressure pain threshold was observed in the painful shoulder of 58 patients with experimental pain response in the shoulder.

In a meta-analysis of patients with shoulder pain, a decrease in pressure pain threshold was found in 29-77% of patients, while SS was found in 11-24% of patients. The authors emphasized the significant correlation of CS with poor treatment response. There is increasing evidence that CS negatively affects various pain treatment responses, including surgery. Considering the frequency of CS in patients with shoulder pain, it is likely to have a negative impact on treatment response in these patients as well. One of the most common treatments for SIS is subacromial/ intra-articular shoulder injection. Although several factors have been identified in the prediction of shoulder injection outcomes, the effect of pain sensitization on these procedures is not yet known.

This study was designed as a prospective single-center study. Patients aged 18-65 years with rotator cuff lesions lasting more than three months and presenting to our physical medicine and rehabilitation outpatient clinic will be included. Patients who have received medical treatment as part of routine practice and have not had an adequate response will be evaluated before and after injection. Injection preference will be determined according to the patient primary complaint and lesion and will be administered into the subacromial space or into the shoulder joint. There is no additional interventional procedure due to the study. Patients will be divided into 2 groups with and without central sensitization. A total of 18 patients were planned for each group. The study will be conducted between March 2023 and June 2024.

Within the scope of the study, age, gender, body mass index, marital status, education level and occupation of the participants will be recorded as demographic data. Clinical evaluation includes pain duration, treatments received, pain intensity (numeric pain scale 0-10), disease-related MRI/USG findings and the following evaluations.

All patients will be evaluated before injection, 1 week, 1 and 3 months after injection. Within the scope of evaluation, Central Sensitization Scale, Quick DASH, SF-36 and Hospital Anxiety and Depression questionnaire, pressure pain threshold, goniometric shoulder range of motion measurement, hand grip strength (with Jamar hydraulic hand dynamometer), numeric pain scale (no pain: 0- unbearable pain: 10) and pain intensity will be recorded at each visit.

Data analysis will be performed by using the Statistical Package for the Social Sciences (SPSS, version 23.0, IBM Corp., Armonk, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

* Clinically and radiographically confirmed rotator cuff pathology
* Being between the ages of 18-65
* Non-response to medical treatment
* Being literate
* To agree to participate in the study

Exclusion Criteria:

* History of shoulder trauma and previous shoulder surgery
* Injection in the shoulder area in the last 3 months
* History of active cancer, systemic inflammatory disease and infection
* Pregnancy
* Under 18 and over 65 years of age
* Illiteracy
* Refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rotator cuff lesion patients aged between 18-65 years old, who have received medical treatment as part of routine practice and have not had an adequate response will be evaluated before and after injection visiting our physical medicine and rehabilitation outpatient clinic between March 2023 and June 2024.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Central Sensitization Scale | 12 months
  The central sensitization scale was developed primarily to detect central sensitization findings in patients with chronic pain and consists of two parts, A and B. In part A, 25 somatic and psychosocial symptoms frequently found in patients with central sensitization are questioned. In part B, the presence of diseases with a well-defined relationship with central sensitization is questioned without participating in the scoring. Patients who score 40 points or more out of a total of 100 points are considered to have central sensitization. Düzce et al. stated that the Central Sensitization Scale can be used as a valid method in the Turkish population to screen the presence of central sensitization in patients presenting with chronic pain.

SECONDARY OUTCOMES:
Range of Motion of Shoulde Joint | 12 months
  Goniometric measurements will be made for both upper extremities. Flexion, extension, abduction, adduction, internal and external rotation angles of the shoulder complex will be evaluated in the measurement.
Hand Grip Test | 12 months
  The purpose of this test is to test the maximum isometric contraction strength of the hand and forearm muscles. A hand grip dynamometer (Jamar) will be used for the test. While the patient is sitting in the chair, the elbows will be close to the body and at 90 degree flexion, the wrist will be in a neutral position. The patient will be asked to grasp the dynamometer and squeeze it as hard as she can, and the average of 3 measurements made with an interval of 10 seconds. The test will be repeated for both upper extremities separately.
Numeric Rating Scale | 12 months
  Shoulder pain, feeling of tension and heaviness on the affected arm will be evaluated separately by numerical scale.
Pain-Pressure Threshold Measurement With an Algometer | 12 months
  The measurement will be performed 2 times with 3 min intervals for each region and the average of these applications will be recorded. Before the test, a trial test will be applied to the patient. With the pressure algometer, pressure will be applied to the selected points until it causes pain and the test will be terminated for that region when the patient feels pain. The measurement includes bilateral shoulder region and left forearm as control region and Wagner manual pressure algometer (1 cm2 probe-10 kg/20 lb) will be used. The selected points will be: 1. Bilateral supraspinatus muscle: 1 cm cranial to the midpoint of the spina scapulae 2. Bilateral infraspinatus muscle: Medial edge of the scapula, intersection of the spina scapula and the inferior scapular angle 3. Bilateral upper trapezius muscle: MidN point of the line joining the acromion and C7 spinous process 4. Left forearm volar face center as control point
Quick Disabilities of the Arm, Shoulder and Hand (Quick DASH) | 12 months
  The arm, shoulder and hand problems rapid questionnaire is a shortened version of a questionnaire designed to detect symptoms and loss of function secondary to musculoskeletal problems of the upper extremity. The questionnaire will be used to assess quality of life related to upper extremity function.
Short Form-36 | 12 months
  The scale was developed by Ware in 1987 and consists of 36 questions in which 8 sub-parameters related to the health status of the person are questioned. These parameters are physical function, pain, limitation due to physical and emotional problems, emotional well-being, social function, fatigue and general health perception. The Turkish validity and reliability of the scale was performed by Pınar et al. It is one of the leading methods used in the evaluation of quality of life in our country as well as all over the world.
Hospital Anxiety and Depression Scale | 12 months
  This scale was developed by Zigmond and Snaith in 1983 to screen anxiety and depression in individuals with physical illness. The scale consists of fourteen questions, seven for anxiety and seven for depression, to be answered on a four-point Likert scale. The Turkish validity and reliability of the scale has been demonstrated and a score above ten for anxiety and seven for depression is considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Ata, Ass. Prof., Principal Investigator — Sultan 2. Abdulhamid Han Training and Research Hospital
Locations (1):
- Sultan 2. Abdulhamid Han Training and Research Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Duzce Keles E, Birtane M, Ekuklu G, Kilincer C, Caliyurt O, Tastekin N, Is EE, Ketenci A, Neblett R. Validity and reliability of the Turkish version of the central sensitization inventory. Arch Rheumatol. 2021 Oct 18;36(4):518-526. doi: 10.46497/ArchRheumatol.2022.8665. eCollection 2021 Dec. PMID 35382371
- [Result] Walankar PP, Panhale VP, Patil MM. Psychosocial factors, disability and quality of life in chronic shoulder pain patients with central sensitization. Health Psychol Res. 2020 Oct 1;8(2):8874. doi: 10.4081/hpr.2020.8874. eCollection 2020 Oct 5. PMID 33123644
- [Result] Previtali D, Bordoni V, Filardo G, Marchettini P, Guerra E, Candrian C. High Rate of Pain Sensitization in Musculoskeletal Shoulder Diseases: A Systematic Review and Meta-analysis. Clin J Pain. 2021 Mar 1;37(3):237-248. doi: 10.1097/AJP.0000000000000914. PMID 33399396
- [Result] Coronado RA, Simon CB, Valencia C, George SZ. Experimental pain responses support peripheral and central sensitization in patients with unilateral shoulder pain. Clin J Pain. 2014 Feb;30(2):143-51. doi: 10.1097/AJP.0b013e318287a2a4. PMID 23619203
- [Result] Sanchis MN, Lluch E, Nijs J, Struyf F, Kangasperko M. The role of central sensitization in shoulder pain: A systematic literature review. Semin Arthritis Rheum. 2015 Jun;44(6):710-6. doi: 10.1016/j.semarthrit.2014.11.002. Epub 2014 Nov 13. PMID 25523242